CLINICAL TRIAL: NCT01749410
Title: A Retrospective Study to Evaluate the Effectiveness and Benefit of onabotulinumtoxinA in Patients With Chronic Migraines
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: GMA-BTX-CM-12-491
Record Dates: First submitted 2012-12-12; First posted 2012-12-13 (Estimated); Results first posted 2015-09-10 (Estimated); Last update posted 2015-09-10 (Estimated); Status verified 2015-08

CONDITIONS: Chronic Migraine, Headaches
MeSH Terms: conditions — Headache | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All participants: Previous treatment with onabotulinumtoxinA for Chronic Migraine based on retrospective medical record review.
  Interventions: Biological: onabotulinumtoxinA

INTERVENTIONS:
Biological: onabotulinumtoxinA — Previous treatment with onabotulinumtoxinA for Chronic Migraine.
  Other Names: Botulinum Toxin Type A; BOTOX®

SUMMARY:
This study will evaluate the effectiveness and benefit of treatment with onabotulinumtoxinA in Chronic Migraine patients who have received a minimum of 7 treatment cycles.

ELIGIBILITY:
Inclusion Criteria:

* 15 or more headache days over a 30 day period
* A minimum of 7 treatment cycles with onabotulinumtoxinA

Exclusion Criteria:

* Any treatment cycle dose of onabotulinumtoxinA greater than 200 units

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who previously received at least 7 treatment cycles of onabotulinumtoxinA as Treatment for Chronic Migraine.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2013-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Encinitas, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Participants
Started | 33
Completed | 33
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.97 (11.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Number of Headache Days
Description: The mean number of headache days was counted as the number of headache days occurring during the 30 day period ending with treatment cycle 7. Each treatment cycle was administered approximately every 12 weeks.
Time Frame: Treatment Cycle 7 (approximately 1.5 years)
Population: All subjects who satisfied the inclusion and exclusion criteria
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | All Participants
Number analyzed (Participants) | 33
Days
  Baseline | 19.08 (5.76)
  Change from Baseline at Cycle 7 (approx 1.5 years) | 6.25 (6.76)

ADVERSE EVENTS:
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 4/33
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=33)
Eyelid Ptosis (Eye disorders) | 2
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.